CLINICAL TRIAL: NCT04589299
Title: Randomized, Parallel Study of Subcutaneous Versus Intravenous Immunoglobulin in Treatment-naïve Patients With Chronic Inflammatory Demyelinating Polyneuropathy
Brief Title: Subcutaneous Immunoglobulin in De-novo CIDP (SIDEC)
Acronym: SIDEC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Rigshospitalet, Denmark (Other); Aarhus University Hospital (Other); Odense University Hospital (Other); Aalborg University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUH-2018-100; 2018-003592-34 (EudraCT Number)
Record Dates: First submitted 2020-09-09; First posted 2020-10-19 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: CIDP - Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: Immunoglobulins, Intravenous; Injections, Subcutaneous
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Immunoglobulins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients treated with immunoglobulin intravenously (IVIG) (Active Comparator): Immunoglobulin (PRIVIGEN) intravenously 2 g/kg/4week for 26 weeks. After this 60 weeks of reduction every 12 weeks (90%, 75%, 50%, 25% and 0%).
  Interventions: Biological: Immunoglobulin
- Patients treated with immunoglobulin subcutaneously (SCIG) (Active Comparator): Immunoglobulin (HIZENTRA) subcutaneously 0.54 g/kg/week for 26 weeks. After this 60 weeks of reduction every 12 weeks (90%, 75%, 50%, 25% and 0%).
  Interventions: Biological: Immunoglobulin

INTERVENTIONS:
Biological: Immunoglobulin — Randomization 1:1 to the same total dose of either SCIG or IVIG for 26 weeks of stable dose + 60 weeks of redcution.

SUMMARY:
SIDEC - (Subcutaneous Immunoglobulin in De-novo CIDP) ia a study designed as a randomized, parallel study with an open-label extension phase. The aims are to compare the effect of SCIG and IVIG in 60 treatment-naïve CIDP patients, and to detect the lowest effective dosage for maintenance treatment.

DETAILED DESCRIPTION:
In fase I the patients are followed for 26 weeks on a fixed dose of 0.54 g/kg/week in the SCIG group (total 14 g/kg) and 2 g/kg/4week in the IVIG group (total 14 g/kg). The patients automatically continue in fase II in which treatment is reduced every 12 weeks (90%, 75%, 50%, 25% and 0%) over a course 60 weeks. The patients are evaluated at every visit with overall disability sum score (ODSS), grip strength, medical research council score (MRC-score), INCAT-Sensory Sum Score (ISS), 10-meter-walk test (10-MWT), 6-spot-step test (6-SST), 9-hole-peg test (9-HPT), quality of life (EQ-5D-5L), Fatigue Severity Scale (FSS), Neuropathic Pain Symptom Inventory (NPSI), Rasch built overall disability scale (RODS) and Life Quality Index (LQI) and blood samples.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling EFNS/PNS criteria for definite, probable or pure motor CIDP.
* No previous treatment with IVIG or SCIG.
* Age ≥ 18.
* ODSS ≥ 2 - either (arm/leg): 1/1, 2/0 or 0/2 at the time of inclusion.

Clinical criteria for typical CIDP

* Chronically progressive, stepwise, or recurrent symmetric proximal and distal weakness and sensory dysfunction of all extremities, developing over at least 2 months; cranial nerves may be affected.
* Absent or reduced tendon reflexes in all extremities.

Criteria for pure motor CIDP • Pure motor affection; otherwise as for typical CIDP.

Electrophysiological criteria for CIDP

1. Motor distal latency prolongation ≥50% above ULN in two nerves (excluding median neuropathy at the wrist from carpal tunnel syndrome), or
2. Reduction of motor conduction velocity ≥30% below LLN in two nerves, or
3. Prolongation of F-wave latency ≥30% above ULN in two nerves (≥50% if amplitude of distal negative peak CMAP ≤80% of LLN values), or
4. Absence of F-waves in two nerves of these nerves have distal negative peak CMAP amplitudes ≥20% of LLN + ≥1 other demyelinating parameter in ≥1 other nerve, or
5. Partial motor conduction block: ≥50% amplitude reduction of the proximal negative peak CMAP relative to distal, if distal negative peak CMAP >20% of LLN, in two nerves, or in one nerve + ≥1 other demyelinating parameter in ≥1 other nerve, or
6. Abnormal dispersion (≥30% duration increase between the proximal and distal negative peak CMAP) in ≥2 nerves, or
7. Distal CMAP duration (interval between onset of the first negative peak an return to baseline of the last negative peak) increase in ≥1 nerve (median ≥6.6 ms, ulnar ≥6.7 ms, peroneal ≥7.6 ms, tibial ≥8.8 ms) + ≥1 other demyelinating parameter in ≥1 other nerve

Electrophysiological criteria for probable CIDP

(a) ≥30% amplitude reduction of the proximal negative peak CMAP relative to distal, excluding the posterior tibial nerve, if distal negative peak CMAP ≥20% of LLN, in two nerves, or in one nerve + ≥1 other demyelinating parameter in ≥1 other nerve

Exclusion Criteria:

* Other causes of neuropathy
* Increased risk of thromboembolism
* Pregnancy (Plasma HCG is tested at inclusion in all fertile women)
* Breast feeding
* Malignancy
* Severe medical disease
* Other immune modulating treatment than low dose steroid (prednisolon < 25 mg daily) within the last 6 months prior to inclusion
* Hepatitis B or C or HIV infection (screening at inclusion)
* Known IgA deficiency
* Known allergy to consents in PRIVIGEN or HIZENTRA
* Body weight > 120 kg

After treatment initiation:

* Pregnancy
* Serious medical disease that affects treatment or examinations
* Non-compliance to treatment
* Initiation of other immune modulating therapy
* Unacceptable side effects
* Withdrawal of consent to participate (drop-out)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in disability | Week 0 to 26
  Evaluated with overall disability sum score (ODSS)

SECONDARY OUTCOMES:
Change in grip strength | Week 0 to 26
  Grip strength (JAMAR)
Change in general muscle strength | Week 0 to 26
  MRC-score
Change in sensation | Week 0 to 26
  INCAT-Sensory Sum Score (ISS)
Change in walking performance | Week 0 to 26
  10-meter-walk test (10-MWT)
Change in walking performance and imbalance | Week 0 to 26
  6-spot-step test (6-SST)
Change in dexterity | Week 0 to 26
  9-hole-peg test (9-HPT)
Change in quality of life | Week 0 to 26
  QoL (EQ-5D-5L incl. VAS)
Change in fatigue severity | Week 0 to 26
  Fatigue Severity Scale (FSS)
Change in pain severity | Week 0 to 26
  Neuropathic Pain Symptom Inventory (NPSI)
Change in disability | Week 0 to 26
  Rasch built overall disability scale (RODS)
Change in treatment satisfaction | Week 2 to 26
  Life Quality Index (LQI)
Serum samples | Week 0 to 26
  Plasma IgG Hematology: hemoglobin, reticulocyte count, haptoglobin, bilirubin, plasma haemoglobin, leukocyte count, thrombocyte count.
  Inflammatory biomarkers: sCD163 and neurofilament
Fluctuations in the describing parameters (ODSS and RODS) in both groups (SCIG and IVIG) based on measurement at time points for treatment with IVIG | Week 0 to 26
  Average value of examinations made at week 0, 4 and 20 (prior to IVIG infusion) Average value of examinations made at week 2, 14 and 26 (2 weeks after IVIG infusion)

OTHER OUTCOMES:
The lowest dose of IVIG or SCIG reached during the 60 weeks of reduction (Fase II). | Week 26 to 86
  Monitored on ODSS and the same secondary parameters as in week 0 to 26

CONTACTS AND LOCATIONS:
Overall Officials: Henning Andersen, MD,DMSc,PhD, Principal Investigator — Aarhus University, Aarhus University Hospital
Locations (4):
- Denmark (4):
  - Department of Neurology, Aalborg University Hospital, Aalborg
  - Department of Neurology, Aarhus University Hospital, Aarhus C
  - Department of Neurology, Rigshospitalet, Copenhagen University Hospital, Copenhagen
  - Department of Neurology, Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No